CLINICAL TRIAL: NCT07377214
Title: AquaTherapy and Subsequent Training for 50 Veterans With PTSD - A Feasibility Study
Brief Title: Effect of Aquatic Therapy and Subsequent Training on Veterans With PTSD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AquaTerapi (Other)
Collaborators: Herlev and Gentofte Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 162026
Record Dates: First submitted 2026-01-16; First posted 2026-01-29 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Post Traumatic Stress Disorder
Keywords: PTSD Aquatherapy feasibility study
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: The project is designed as a single-group pre-post feasibility study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aquatic Therapy and subsequent Group Training for Veterans With PTSD: 32-Week Feasibility Study (Experimental): This arm consists of a 32-week intervention for veterans diagnosed with PTSD. The first phase is 16 weeks of individual Aquatic Therapy delivered twice weekly in a 34°C warm water pool by a physiotherapist, focusing on relaxation, movement, and body awareness.
  The second phase is 16 weeks of group-based aquatic training, held once weekly in small groups, emphasizing cardiovascular fitness, strength, mobility, and relaxation. The intervention aims to reduce PTSD symptoms, improve sleep quality, and enhance quality of life. Outcomes are measured before, after, and at one-year follow-up using validated questionnaires (PCL-M, PSQI, WHO-5, HSCL-25) and participant feedback.
  The program is delivered by experienced physiotherapists and is considered safe and non-invasive. The study is conducted in collaboration with military psychiatric services, veteran organizations, and academic partners
  Interventions: Other: AquaTherapy

INTERVENTIONS:
Other: AquaTherapy — The intervention consists of a 32-week program for veterans diagnosed with PTSD, delivered in two consecutive phases. The first phase comprises 16 weeks of individual Aquatic Therapy where each participant receives one-on-one aquatic physiotherapy sessions with a trained physiotherapist in a warm water pool (34-36°C), twice weekly. These sessions focus on relaxation, gentle movement, and body awareness, aiming to reduce stress and establish a sense of safety and calm.
  Following the individual phase, participants transition to a 16-week group-based aquatic training program. This second phase involves weekly sessions in small groups (up to six participants per group) and emphasizes cardiovascular fitness, strength, mobility, and relaxation, all conducted in the same warm water environment. The group format is designed to reinforce physical gains, promote social engagement, and support the maintenance of improved activity levels.
  Other Names: Aquatic group training

SUMMARY:
This project investigates the effect of Aquatic Therapy followed by group training for 50 veterans diagnosed with PTSD.

Around 40% of Danish veterans experience insufficient benefit from current standard treatments, especially regarding sleep and quality of life.

The study is a single-group, pre-post feasibility study, where participants receive 16 weeks of individual aquatic therapy (twice weekly) in a 34 °C pool, followed by 16 weeks of group-based aquatic exercise (once weekly). Participants are recruited through military psychiatric clinics and veteran organizations.

The primary outcome is change in PTSD symptoms measured by the PCL-M questionnaire. Secondary outcomes include sleep quality (PSQI), quality of life (WHO-5), anxiety and depression (HSCL-25), and social participation. Data are collected before, after, and at one-year follow-up. The study also evaluates feasibility in terms of recruitment, adherence, acceptability, and follow-up rates.

The aim is to achieve clinically relevant reductions in PTSD symptoms, improved sleep, and enhanced quality of life. The project is conducted in collaboration with military psychiatric services, and veteran organizations, and is managed by Gentofte Hospital. The intervention is considered safe and non-invasive, and all ethical and data protection regulations are followed. The project will provide rapid access to new treatment, generate knowledge for national implementation. Previous studies indicate marked and lasting improvements in sleep, symptoms, and quality of life, supporting reintegration into work and social life.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) is prevalent among military veterans and is commonly associated with persistent hyperarousal, sleep disturbances, and reduced quality of life. Although trauma-focused psychotherapy and pharmacological treatment are considered first-line interventions, a substantial proportion of veterans continue to experience residual symptoms, particularly related to sleep, physiological stress regulation, and daily functioning. This highlights the need for complementary, non-pharmacological interventions that address both psychological and somatic aspects of PTSD.

Aquatic therapy delivered in warm water represents a body-based intervention with potential relevance for trauma-exposed populations. The physical properties of warm water, including buoyancy, hydrostatic pressure, and thermal effects, may facilitate relaxation, reduce muscle tension, and support autonomic nervous system regulation. Trauma-informed aquatic therapy further emphasizes safety, predictability, and bodily awareness, which are considered central mechanisms in reducing hyperarousal and improving sleep and well-being in individuals with PTSD. Preliminary Danish and international studies suggest that aquatic therapy is safe and may lead to clinically meaningful improvements in PTSD-related symptoms, sleep quality, and quality of life among veterans with chronic PTSD.

The present study evaluates a structured, two-phase aquatic intervention consisting of an initial individual therapy phase followed by group-based aquatic exercise. The individual phase is designed to establish a sense of safety, promote relaxation, and enhance body awareness through one-to-one sessions with a physiotherapist in a warm water environment. This phase aims to reduce physiological stress responses and prepare participants for more active and socially oriented exercise. The subsequent group-based phase focuses on gradual reintroduction of physical activity and social participation through supervised aquatic exercise, with the intention of consolidating treatment gains and supporting longer-term maintenance.

The study is conducted as a single-group, pre-post feasibility study. The primary objective is to assess the feasibility of delivering the intervention to veterans with PTSD, including recruitment procedures, adherence to the intervention, acceptability of the treatment model, and the practicality of follow-up assessments. As a feasibility study, the trial is not powered to test efficacy, but to inform the design, procedures, and outcome selection for a future randomized controlled trial. Secondary objectives include exploring changes in PTSD-related symptoms, sleep quality, and quality of life to support planning of subsequent controlled studies.

Data are collected at baseline, immediately after completion of the intervention, and at one-year follow-up using validated self-report instruments. In addition, qualitative feedback is collected to capture participant experiences, perceived benefits, and potential barriers to participation. These data will be used to refine the intervention protocol and study procedures prior to potential scaling or evaluation in a controlled trial.

The intervention is non-invasive and delivered by experienced physiotherapists trained in aquatic therapy for trauma-exposed populations. All study procedures are conducted in accordance with applicable ethical guidelines and data protection regulations

ELIGIBILITY:
Inclusion Criteria:

* Veteran diagnosed with PTSD.
* Willingness to complete questionnaires and respond to texts.
* Sufficient Danish language proficiency
* Practical ability to participate (sessions are Wednesday and Friday afternoons)
* Able to attend or arrange transport to Tuborgvej, 2400 Copenhagen NV
* Any substance abuse must be under control

Exclusion Criteria:

* Acute psychiatric crisis or severe comorbid psychiatric disorder that would prevent participation.
* Physical conditions that contraindicate participation in aquatic therapy (e.g., open wounds, severe infections, or other medical contraindications for warm water therapy).
* Lack of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in PTSD symptoms measured by the PTSD Checklist - Military Version (PCL-M) | Baseline, end of 32-week intervention, and 1-year follow-up.
  Outcome Measure Description: Change in PTSD symptom severity assessed using the Posttraumatic Stress Disorder Checklist - Military Version (PCL-M). The PCL-M is a 17-item self-report questionnaire with total scores ranging from 17 to 85, where higher scores indicate more severe PTSD symptoms. A clinically meaningful improvement is defined as a reduction of ≥10 points from baseline.

SECONDARY OUTCOMES:
Change in sleep quality measured by the Pittsburgh Sleep Quality Index (PSQI) | Baseline, end of 32-week intervention, and 1-year follow-up.
  Outcome Measure Description: Change in sleep quality assessed using the Pittsburgh Sleep Quality Index (PSQI). The PSQI global score ranges from 0 to 21, where higher scores indicate poorer sleep quality. Clinically relevant improvement is defined as a reduction of ≥3 points in the global score or achieving a score of ≤5.
Change in quality of life measured by the WHO-5 Well-Being Index | Baseline, end of 32-week intervention, and 1-year follow-up.
  Change in psychological well-being assessed using the World Health Organization-Five Well-Being Index (WHO-5). Scores range from 0 to 100, where higher scores indicate better well-being and quality of life. A change of ≥10 points is considered clinically meaningful.

OTHER OUTCOMES:
Change in anxiety and depression symptoms measured by the Hopkins Symptom Checklist-25 (HSCL-25) | Baseline, end of 32-week intervention, and 1-year follow-up.
  Change in anxiety and depression symptom severity assessed using the Hopkins Symptom Checklist-25 (HSCL-25). The mean score ranges from 1.0 to 4.0, where higher scores indicate greater symptom severity. A commonly used clinical cut-off is 1.75.
Feasibility measure: Adherence Rate | End of intervention (week 32).
  Proportion of enrolled participants who complete the full intervention program. Higher values indicate better adherence.
Feasibility measure: Acceptability | End of intervention (week 32).
  Proportion of participants who report that they would recommend the intervention to other veterans with PTSD. Higher values indicate greater acceptability.
Feasibility measure: 1-Year Follow-Up Rate | End of intervention (week 32).
  Proportion of participants who complete the 1-year follow-up assessment. Higher values indicate better retention.
Feasibility measure: Recruitment Rate | End of intervention (week 32).
  Proportion of the planned sample size that is successfully recruited and enrolled within the predefined recruitment period. Higher values indicate better recruitment feasibility.
Explorative outcome: Weekly Visual Analogue Scale (VAS) Scores | Weekly during the 32-week intervention period.
  Weekly self-reported ratings using Visual Analogue Scales (VAS) ranging from 0 to 10. Higher scores indicate greater intensity or frequency of the rated domain (e.g., intrusive thoughts, calmness, self-esteem, sleep quality, physical activity, mood).
Explorative outcome: Qualitative Interviews | End of intervention (week 32) and 1-year follow-up.
  Semi-structured qualitative interviews exploring participant experiences, perceived changes in daily functioning, and overall satisfaction with the intervention. Data are analyzed thematically.
Explorative outcome: Open-Ended Participant Feedback | End of intervention (week 32).
  Written open-ended feedback collected to explore perceived benefits, barriers, and acceptability of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Bogh Juhl, Prof., Principal Investigator — Herlev & Gentofte Hospital
Locations (1):
- AquaTerapi, Tuborgvej, 2400 Copenhagen NV, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website presenting our research and clinical experience with Aquatic Therapy for stress and PTSD — http://www.aquaterapi.dk